CLINICAL TRIAL: NCT01146899
Title: FluAlert: Influenza Vaccine Alerts for Providers in the Electronic Health Record
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Asst Prof of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAE4956; 1R18HS018158-01 (AHRQ)
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Influenza
Keywords: influenza, vaccine, clinical decision support
MeSH Terms: conditions — Influenza, Human | interventions — Caffeine; Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provider Alert (Experimental): Provider receives alert for patient visit
  Interventions: Other: Provider Alert
- No Alert (No Intervention): No alert provided

INTERVENTIONS:
Other: Provider Alert — Provider influenza vaccine alert
  Other Names: alert for provider in electronic health record
  Arms: Provider Alert

SUMMARY:
Childhood influenza coverage rates are far below rates for the other childhood vaccinations. Increasing influenza vaccine coverage rates is important not only for the health of the child, but for that of the child's household and community. Yet,influenza vaccine delivery rates at pediatric clinics are low, even when the vaccine is available. The proposed project will take advantage of existing health information technology to tailor, implement and evaluate influenza vaccine alerts in the electronic health record (EHR) for pediatric providers to help improve health care decision making.

ELIGIBILITY:
Inclusion Criteria:

* Medical (medical doctor/nurse practitioner (MD/NP)) or nursing providers (registered nurse, licensed practical nurse (RN/LPN)) at participating practices
* Parents of a child 6 months - 18 years who is a patient at one of the participating ACN practice
* Parents fluent in English or Spanish
* Children 6 months- 18 years with visit to participating practice during influenza season

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6145 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
influenza vaccination | September through March 2011-2012

SECONDARY OUTCOMES:
Documentation of reason for vaccine refusal | Sept 2011-March 2012

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center/ NewYork Presbyterian Hospital Ambulatory Care Network, New York, New York, United States

REFERENCES:
- [Derived] Stockwell MS, Catallozzi M, Camargo S, Ramakrishnan R, Holleran S, Findley SE, Kukafka R, Hofstetter AM, Fernandez N, Vawdrey DK. Registry-linked electronic influenza vaccine provider reminders: a cluster-crossover trial. Pediatrics. 2015 Jan;135(1):e75-82. doi: 10.1542/peds.2014-2616. PMID 25548331